CLINICAL TRIAL: NCT00936936
Title: High-dose Chemotherapy for Poor-Prognosis Relapsed Germ-Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0378; NCI-2011-01631 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Testicular Cancer
Keywords: Testis; Relapsed Testicular Cancer; Bevacizumab; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Carboplatin; Paraplatin; Docetaxel; Taxotere; Etoposide; VePesid; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Ifosfamide; Ifex; Melphalan; Alkeran
MeSH Terms: conditions — Testicular Neoplasms | interventions — Gemcitabine; Docetaxel; Melphalan; Carboplatin; Mesna; Ifosfamide; Etoposide; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cycle # 1 (Experimental): First Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  HD Cycle #1: Gemcitabine/Docetaxel/Melphalan/Carboplatin + PBPC
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Melphalan; Drug: Carboplatin; Procedure: Stem Cell Transplant
- Cycle #2 (Experimental): Second Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  HD Cycle #2: Ifosfamide/Carboplatin/Etoposide + PBPC
  Interventions: Drug: Carboplatin; Drug: Mesna; Drug: Ifosfamide; Drug: Etoposide; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Gemcitabine — 1800 mg/m^2 IV over 3 hours on Days -5 to Day -2.
  Other Names: Gemcitabine Hydrochloride; Gemzar
  Arms: Cycle # 1
Drug: Docetaxel — Docetaxel 300 mg/m^2 IV over 2 hours on Day -5.
  Other Names: Taxotere
  Arms: Cycle # 1
Drug: Melphalan — 50 mg/m^2 IV over 15 minutes on Days -4 to Day -2.
  Other Names: Alkeran
  Arms: Cycle # 1
Drug: Carboplatin — Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Cycle #2: 300 mg/m^2 IV over 2 hours on Days -6 to -3.
  Other Names: Paraplatin
Drug: Mesna — 3,000 mg/m^2 per day in 96-hour continuous infusion, starting 30 minutes prior to the first dose of ifosfamide, on Days -6 to -4.
  Other Names: Mesnex
  Arms: Cycle #2
Drug: Ifosfamide — 3,000 mg/m^2 IV over 6 hours on Days -6 to -3
  Other Names: Ifex
  Arms: Cycle #2
Drug: Etoposide — 200 mg/m^2 IV over 3 hours, every 12 hours on Days -6 to -4.
  Other Names: VePesid
  Arms: Cycle #2
Procedure: Stem Cell Transplant — Stem cell infusion on Day 0.
  Other Names: SCT; Hematopoietic progenitor-cell infusion; PBPC

SUMMARY:
The goal of this clinical research study is to learn if 2 cycles of high-dose chemotherapy can help to control germ-cell tumors. The first cycle of chemotherapy will include the drugs gemcitabine, docetaxel, melphalan, and carboplatin. The second cycle of chemotherapy will include the drugs ifosfamide, carboplatin, and etoposide. The safety of these drug combinations will also be studied.

This is an investigational study. Gemcitabine, docetaxel, melphalan, ifosfamide, carboplatin, and etoposide are all FDA-approved and commercially available for the treatment of germ-cell tumors.

Up to 67 patients will be enrolled in this study.

DETAILED DESCRIPTION:
The Study Drugs:

Carboplatin, melphalan, and ifosfamide are designed to damage the DNA (the genetic material) of cancer cells, which may cause the cancer cells to die.

Docetaxel and etoposide are designed to stop the growth of cancer cells, which may cause the cancer cells to die.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die. It may also help docetaxel, carboplatin, and melphalan to be more effective by stopping tumor cells from repairing damage caused by these drugs.

Study Drug Administration:

You will receive 2 cycles of high-dose chemotherapy with stem-cell support, 1-2 months apart.

You will receive 1 dose of Outpatient IV at Bevacizumab 7.5mg/kg.

Starting on the first day of your hospital stay, you will begin gargling and swishing Caphosol and Glutamine in your mouth 4 times a day. This is done to help prevent mouth and throat sores.

On Day 2 of your stay in the hospital, through the CVC, you will receive gemcitabine over 4 hours and docetaxel over 2 hours.

On Days 3-5, through the CVC, you will receive gemcitabine over 4 hours, melphalan over 15 minutes, and carboplatin over 2 hours.

On Day 6, you will not receive any study drugs.

On Day 7, you will receive the stem cells through the CVC over about 30-60 minutes.

As part of standard care, you will receive G-CSF (filgrastim) as an injection under your skin daily, starting 5 days after the transplant, until your blood cell levels return to normal.

As part of standard mouth care you will be asked to do mouthwashes 4 times a day with caphosol (artificial saliva) and glutamine.

Two (2) to 4 weeks after you leave the hospital after Cycle 1, you will receive your second cycle of high-dose chemotherapy.

On Days 2-4 of your stay in the hospital, through the CVC, you will receive ifosfamide over 6 hours, etoposide over 2 hours, and carboplatin over 2 hours.

On Days 5-6, you will not receive any study drugs.

On Day 7, you will receive the stem cells through the CVC over about 30-60 minutes.

Study Visits:

About 1 month, 100 days, 6 months and 1 year after your second stem cell transplant, the following tests and procedures will be performed:

* To check the status of the disease, you will have CT scans of your chest, abdomen, and pelvis.
* Blood (about 3 tablespoons) will be drawn for routine tests.

Length of Study:

You will be off study after about 1 year from your second transplant. You will be taken off study early if the disease gets worse or if you experience any intolerable side effects.

Long-Term Follow-up:

If your doctor thinks it is needed, you may have follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age 12 to 65 years.
2. Patients with seminomatous or nonseminomatous germ-cell tumors (GCT) in one of the following groups: A) First relapse or progression or second response with an intermediate or high risk according to the Beyer model. B) Second relapse or beyond.
3. Adequate renal glomerular and tubular function, as defined by estimated serum creatinine clearance >/=50 ml/min and/or serum creatinine </= 1.8 mg/dL, and urinary protein excretion </=500 mg/day.
4. Adequate hepatic function, as defined by ALT and AST </=3 x upper limit of normal (ULN); serum bilirubin and alkaline phosphatase </=2 x ULN or considered not clinically significant.
5. Adequate pulmonary function with FEV1 (Forced expiratory volume in the first second), FVC (Forced vital capacity) and DLCO (diffusing capacity of the lung for carbon monoxide) >/=50% of predicted, corrected for volume and hemoglobin.
6. Adequate cardiac function with LVEF (left ventricular ejection fraction) >/=40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
7. Zubrod performance status 0-2.
8. A minimum apheresis collection of 5 million CD34+ cells/kg of autologous hematopoietic progenitor cells (AHPC).
9. Written informed consent by patients and/ or their parents or legal guardians. Assent for those patients inclusive of ages 12 to 17.

Exclusion Criteria:

1. Growing teratoma syndrome, defined as enlarging tumor masses with normal serum markers during chemotherapy for nonseminomatous GCT.
2. Major surgery within 30 days before the initiation of study treatment
3. Radiotherapy within 21 days prior to initiation of study treatment
4. Prior whole brain irradiation.
5. Patients with active central nervous system (CNS) disease, defined as brain or meningeal metastases that are not in complete remission.
6. Patients with active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA >/=10,000 copies/mL, or >/= 2,000 IU/mL).
7. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients who either show chronic hepatitis C or positive hepatitis C serology.
8. Active infection requiring parenteral antibiotics.
9. HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal CD4 counts
10. Patients who have had a previous autologous or allogeneic stem cell transplant in the previous 12 months.
11. Positive pregnancy test in a female patient of childbearing potential defined as not post menopausal for twelve months or no previous surgical sterilization.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-06-02 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PHD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Nieto Y, Tu SM, Bassett R, Jones RB, Gulbis AM, Tannir N, Kingham A, Ledesma C, Margolin K, Holmberg L, Champlin R, Pagliaro L. Bevacizumab/high-dose chemotherapy with autologous stem-cell transplant for poor-risk relapsed or refractory germ-cell tumors. Ann Oncol. 2015 Oct;26(10):2125-32. doi: 10.1093/annonc/mdv310. Epub 2015 Jul 21. PMID 26199392
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer Center.
Groups:
- Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT: First Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  You will receive 1 dose of Outpatient IV at Bevacizumab 7.5mg/kg.
  HD Cycle #1: Gemcitabine/Docetaxel/Melphalan/Carboplatin + PBPC
  Gemcitabine: 1800 mg/m^2 IV over 3 hours on Days -5 to Day -2.
  Docetaxel: Docetaxel 300 mg/m^2 IV over 2 hours on Day -5.
  Melphalan: 50 mg/m^2 IV over 15 minutes on Days -4 to Day -2.
  Carboplatin: Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Stem Cell Transplant: Stem cell infusion on Day 0.
  Second Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  HD Cycle #2: Ifosfamide/Carboplatin/Etoposide (ICE) + PBPC
  Carboplatin: Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Cycle #2: 300 mg/m^2 IV over 2 hours on Days -6 to -3.
  Mesna: 3,000 mg/m^2 per day in 96-hour continuous infusion, starting 30 minutes prior to the first dose of ifosfamide, on Days -6 to -4.
  Ifosfamide: 3,000 mg/m^2 IV over 6 hours on Days -6 to -3
  Etoposide: 200 mg/m^2 IV over 3 hours, every 12 hours on Days -6 to -4.
  Stem Cell Transplant: Stem cell infusion on Day 0.
- Cohort 2: HD GeM-DMC+ ICE for Refractory GCT: First Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  HD Cycle #1: Gemcitabine/Docetaxel/Melphalan/Carboplatin + PBPC
  Gemcitabine: 1800 mg/m^2 IV over 3 hours on Days -5 to Day -2.
  Docetaxel: Docetaxel 300 mg/m^2 IV over 2 hours on Day -5.
  Melphalan: 50 mg/m^2 IV over 15 minutes on Days -4 to Day -2.
  Carboplatin: Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Stem Cell Transplant: Stem cell infusion on Day 0.
  Second Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  HD Cycle #2: Ifosfamide/Carboplatin/Etoposide + PBPC
  Carboplatin: Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Cycle #2: 300 mg/m^2 IV over 2 hours on Days -6 to -3.
  Mesna: 3,000 mg/m^2 per day in 96-hour continuous infusion, starting 30 minutes prior to the first dose of ifosfamide, on Days -6 to -4.
  Ifosfamide: 3,000 mg/m^2 IV over 6 hours on Days -6 to -3
  Etoposide: 200 mg/m^2 IV over 3 hours, every 12 hours on Days -6 to -4.
  Stem Cell Transplant: Stem cell infusion on Day 0.
Period: Overall Study
Arm/Group | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT
Started | 41 | 23
Cycle 1 | 41 | 23
Cycle 2 | 29 | 23
Completed | 29 | 19
Not Completed | 12 | 4
Not completed — Adverse Event | 7 | 1
Not completed — Disease Progression | 2 | 2
Not completed — Unrelated | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT: First Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  You will receive 1 dose of Outpatient IV at Bevacizumab 7.5mg/kg.
  HD Cycle #1: Gemcitabine/Docetaxel/Melphalan/Carboplatin + PBPC
  Gemcitabine: 1800 mg/m^2 IV over 3 hours on Days -5 to Day -2.
  Docetaxel: Docetaxel 300 mg/m^2 IV over 2 hours on Day -5.
  Melphalan: 50 mg/m^2 IV over 15 minutes on Days -4 to Day -2.
  Carboplatin: Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Stem Cell Transplant: Stem cell infusion on Day 0.
  Second Cycle High-dose (HD) chemotherapy followed by stem-cell infusion (PBPC)
  HD Cycle #2: Ifosfamide/Carboplatin/Etoposide + PBPC
  Carboplatin: Cycle 1: 333 mg/m^2 IV over 2 hours on Days -4 to -2.
  Cycle #2: 300 mg/m^2 IV over 2 hours on Days -6 to -3.
  Mesna: 3,000 mg/m^2 per day in 96-hour continuous infusion, starting 30 minutes prior to the first dose of ifosfamide, on Days -6 to -4.
  Ifosfamide: 3,000 mg/m^2 IV over 6 hours on Days -6 to -3
  Etoposide: 200 mg/m^2 IV over 3 hours, every 12 hours on Days -6 to -4.
  Stem Cell Transplant: Stem cell infusion on Day 0.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT | Total
Number analyzed (Participants) | 41 | 23 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 39 | 22 | 61
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 38 | 21 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 20 | 11 | 31
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 41 | 23 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 2-year Event-Free Survival (EFS)
Description: Event-free survival estimated from the first day of High-Dose Course Cycle #1 (Day -6) until tumor progression, relapse, or death from any cause.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT
Number analyzed (Participants) | 41 | 23
Participants | 28 | 11

2. Secondary Outcome: Overall Survival
Description: Number of Participants alive and disease free 1 year post treatment completion.
Time Frame: 1 year post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT
Number analyzed (Participants) | 41 | 23
Participants | 25 | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT
All-Cause Mortality (participants affected / at risk) | 22/41 | 12/23
Serious Adverse Events (participants affected / at risk) | 7/41 | 2/23
Other Adverse Events (participants affected / at risk) | 41/41 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT (N=41) | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT (N=23)
ALT increased (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
Bacterial (Infections and infestations) | 7 (7) | 0 (0)
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Ejection fraction decreased (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 2 (2)
Fungal (Infections and infestations) | 6 (6) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Viral (Infections and infestations) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DAH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HD GeM-DMC+ ICE + Bevacizumab for Refractory GCT (N=41) | Cohort 2: HD GeM-DMC+ ICE for Refractory GCT (N=23)
ALK increased (Investigations) | 4 (4) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
ALT increased (Investigations) | 41 (70) | 22 (22)
AST increased (Investigations) | 6 (6) | 2 (2)
Bacterial (Infections and infestations) | 37 (37) | 14 (14)
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 38 (63) | 23 (32)
Dysrhythmia (Cardiac disorders) | 9 (9) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 5 (5) | 3 (3)
Creatinine increased (Investigations) | 27 (27) | 16 (16)
Diarrhea (Gastrointestinal disorders) | 38 (39) | 14 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ejection fraction decreased (Cardiac disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 35 (35) | 1 (1)
Flu like syndrome (General disorders) | 1 (1) | 1 (1)
Fluid overload (General disorders) | 38 (58) | 23 (23)
Fungal (Infections and infestations) | 14 (14) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 38 (87) | 23 (35)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Lower Gl track obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 38 (78) | 23 (41)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
GI OTH (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Hemorrhagic Cystitis (Renal and urinary disorders) | 3 (3) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 26 (26) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
T bilirubin increased (Investigations) | 36 (36) | 13 (13)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 5 (5) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 38 (47) | 4 (4)
renal failure & fluid retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 0 (0)
SK DES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin Disorders (Skin and subcutaneous tissue disorders) | 38 (63) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Viral (Infections and infestations) | 16 (16) | 5 (5)
DAH (General disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT00936936/Prot_SAP_000.pdf